CLINICAL TRIAL: NCT06314633
Title: Socioeconomic Determinants of the Chemical Exposome and Its Genotoxic Effects in Children
Acronym: PESTIFOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: ANSES (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ICO-2023-13
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer Children
Keywords: DNA damage; Chemical exposome; Hair polluants impregnations; Socio-economic characteristics

STUDY DESIGN:
Intervention Model Description: Hair collection and parents questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study procedures (Other): Hair cut for DNA damage and chemical exposome variation analysis and Socio-economic characteristics
  Interventions: Other: Hair cut; Other: Socio-economic questionnaires

INTERVENTIONS:
Other: Hair cut — Hair locks and follicles will be cut twice in winter and spring
Other: Socio-economic questionnaires — Information about parents education levels and professional occupation, geographic area, children gender, indoor and outdoor children's environmental exposures

SUMMARY:
PESTIFOL will include children over 8 and under 12 years old of different socioeconomic positions (SEP), mostly living in the region of Pays de la Loire. This approach should enable us to assess the impact of the SEP, and therefore social inequalities, on chemical expositions and DNA damage, and to characterize which (classes/mixture of) pollutants are major source of DNA damage. The study will also address potential effects associated with geographical location on the exposome and its biological consequences.

DETAILED DESCRIPTION:
Growing evidence points to a complex influence of the exposome on health outcomes. Epidemiological studies show associations between pesticides and cognitive delay and cancers. Only few were conducted in children. Chemical exposures differ between socioeconomic groups. The more disadvantaged the group, the higher are some exposures. However, the effect of the exposome on health is complicated to assess due to the long latencies of most diseases. It is therefore important to link social and chemical exposures to 'immediate' outcomes or molecular risk factors for human diseases. There is a strong connection between DNA damage and chronic diseases such as cancers. However, it is difficult to attribute these risks to specific impregnations.

The present study will address the impact of socioeconomic position, hence social inequalities, on environmental exposures and their biological consequences in children. Our approach is to detect DNA damage in hair follicles and associate these measurements with pesticide detections in the hair matrix and socioeconomic position (SEP).

PESTIFOL will include children over 8 and under 12 years old of different socioeconomic positions (SEP), mostly living in the region of Pays de la Loire. This approach should enable us to assess the impact of the SEP, and therefore social inequalities, on chemical expositions and DNA damage, and to characterize which (classes/mixture of) pollutants are major source of DNA damage. The study will also address potential effects associated with geographical location on the exposome and its biological consequences.

ELIGIBILITY:
Inclusion Criteria:

* Children over 8 and under 12 years old at the time of inclusion
* Children in school in class level CE2, CM1 or CM2
* Living in the Pays de La Loire region, at least 80% of the time
* Written informed assent and consent obtained from the participant and both parents or legal representative prior to performing any protocol-related procedures.

Exclusion Criteria:

- Disorder precluding understanding of trial information or informed assent.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Describe DNA damage | 4-6 months
  Hair locks and hair follicles will be collected and will be analysed to evaluate the DNA damage : average amount of DNA break foci per nucleus cross-section
Describe DNA damage | 4-6 months
  Hair locks and hair follicles will be collected and will be analysed to evaluate the DNA damage: proportion of cells with an abnormal break rate.
Describe socio-economic characteristics. | 4-6 months
  The socio-economic characteristics will evaluated via parent's questionnaires : parents occupation and education level
Describe socio-economic characteristics. | 4-6 months
  The socio-economic characteristics will evaluated via parents questionnaires : parents education level

SECONDARY OUTCOMES:
Characterize chemical exposome variations | 4-6 months
  Chemical exposome: presence and amount of pollutant impregnations : total number of polluants detected in hair sample
Characterize chemical exposome variations | 4-6 months
  Chemical exposome: presence of pollutants/pesticides classified as genotoxic/carcinogenic by the WHO IARC (International Agency for Research on Cancer), and/or the US EPA (National Environmental Protection Agency).
Characterize socio-economic indicators | 4-6 months
  The socio-economic characteristics will be evaluated via parents' questionnaires: parents' occupation and education level
Characterize socio-economic indicators, geographical area, seasons | 4-6 months
  The socio-economic characteristics will be evaluated via parents' questionnaires: geographic area
Characterize socio-economic indicators, geographical area, seasons | 4-6 months
  The socio-economic characteristics will be evaluated via parents' questionnaires: gender
Characterize socio-economic indicators, geographical area, seasons | 4-6 months
  The socio-economic characteristics will be evaluated via parents' questionnaires: seasons (winter and spring)
Describe DNA damage | 4-6 months
  Evaluate the DNA damage: average amount of DNA break foci per nucleus cross-section
Describe DNA damage | 4-6 months
  Evaluate the DNA damage: proportion of cells with an abnormal break rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancérologie de l'ouest, Saint-Herblain, France